CLINICAL TRIAL: NCT00900887
Title: Efficacy of Topic Antiinflammatory Therapy Treatment in Center Point Thickness Secondary to Selective Photocoagulation in Diabetic Macular Edema
Brief Title: Topic Antiinflammatory Therapy Added to Selective Photocoagulation in Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Juarez de Mexico (Other Government)
Responsible Party: Principal Investigator, Virgilio Lima Gomez, PhD, Hospital Juarez de Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HJM 1470/08.03.18
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Diabetic Retinopathy; Macular Edema
Keywords: diabetic retinopathy; clinically significant macular edema; selective photocoagulation; topic ketorolac; topic nepafenac; efficacy; treatment
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema | interventions — Ketorolac; nepafenac

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ketorolac (Active Comparator): ocular topic ketorolac used 3 times a day for a week after the selective photocoagulation
  Interventions: Drug: Ketorolac
- Nepafenac (Active Comparator): ocular topic nepafenac 3 times a day during one week after selective photocoagulation
  Interventions: Drug: Nepafenac
- Polietilenglicol 400, propilenglicol (Placebo Comparator): ocular lubricant drops 3 times a day for a week after selective photocoagulation
  Interventions: Drug: Polietilenglicol 400, propilenglicol

INTERVENTIONS:
Drug: Ketorolac — ophthalmic presentation 5 mg/ml dosage one drop (0.25 mg) in the treated eye 3 times a day during one week
  Other Names: Godek
  Arms: Ketorolac
Drug: Nepafenac — topic presentation 1 mg/ml dosage one drop (0.05 mg) in the treated eye 3 times a day during one week
  Other Names: Nevanac
  Arms: Nepafenac
Drug: Polietilenglicol 400, propilenglicol — ocular presentation Polietilenglicol 400 (4 mg), propilenglicol (3 mg), HP guar (1.9 mg)/1 ml
  dosage: one drop (0.2 mg polietinglicol 400, 0.15 mg propilenglicol, 0.095 mg HP guar) 3 times a day during one week
  Other Names: Systane
  Arms: Polietilenglicol 400, propilenglicol

SUMMARY:
The purpose of this study is to determine the efficacy of ocular topic antiinflammatory therapy (sodic nepafenac at 0.1% or ketorolac at 0.5%) to treat center point thickness secondary to selective photocoagulation in diabetics with clinically significant macular edema.

DETAILED DESCRIPTION:
Selective photocoagulation is the standard treatment for clinically significant macular edema. This treatment decreased the incidence of moderate visual loss in the long term. Nonetheless, in the first six weeks after treatment it is induced, probably because an exacerbation of macular edema secondary to treatment. An inflammatory response has been reported after selective photocoagulation. Therefore, antiinflammatory therapy like ketorolac or nepafenac could be useful to manage center point thickness secondary to selective photocoagulation in diabetics with macular edema.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* regardless of diabetes duration and retinopathy severity level
* one or both eyes with focal clinically significant macular edema
* treated with selective or focal photocoagulation
* visual capacity under subjective refraction before treatment
* adequate quality 6mm fast macular map on the day of photocoagulation
* signed of inform consent

Exclusion Criteria:

* ocular surgery in the last 4 months
* previous selective photocoagulation
* topic or systemic antiinflammatory therapy in the last week
* allergic to antiinflammatory non-steroids therapy
* lent contact used in tha last 2 days before photocoagulation
* history of ocular trauma, ocular infection or lacrimal dysfunction in the last 3 months
* history of uveitis or ocular inflammation in the last 12 months
* any ocular external disease, infection or inflammatory process during evaluation
* corneal abnormalities that could modify visual capacity per se
* actual corneal disease
* pregnancy
* myopia over -6.00 diopters
* any retinal disease different from diabetic retinopathy
* adverse event of the drug
* desert to pharmacology therapy after the second visit
* no assistance after the second visit
* inadequate quality 6mm fast macular map after the second visit

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2008-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
ocular topic antiinflammatory therapy (ketorolac, nepafenac or placebo) applied 3 times a day in the treated eye for a week after selective photocoagulation | one week after treatment

SECONDARY OUTCOMES:
center point thickness using stratus OCT measured in microns | before treatment, at 24, 48 and 168 hours after treatment
macular volume using stratus OCT measured in cubic millimeters | before treatment, 24, 48 and 168 hours after treatment
visual capacity under subjective refractive correction measured in decimal equivalent | before treatment, at 24, 48, 168 hours after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Virgilio Lima Gomez, MD, MSc, Study Chair — Hospital Juarez de Mexico; Dulce M Razo Blanco Hernandez, MD, Principal Investigator — Hospital Juarez de Mexico; Juan Asbun Bojalil, MD, PhD, Study Director — Hospital Juarez de Mexico
Locations (1):
- Virgilio Lima Gomez, Mexico City, Mexico City, Mexico